CLINICAL TRIAL: NCT00616928
Title: A Trial to Evaluate the Safety and Immunogenicity of an Investigational Vaccination Regimen in Adults Aged ≥18 Years
Brief Title: Immunogenicity & Safety of GSK's Influenza Vaccine 1557484A Given to Adults Aged ≥18 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 110464
Record Dates: First submitted 2008-01-28; First posted 2008-02-15 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: vaccines; immunogenicity; human; safety; influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (10):
- Influenza A (H5N1) 18-64Y Group (Experimental): Subjects aged 18-64 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted vaccine formulations A. B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted
- Placebo 18-64Y Group (Placebo Comparator): Subjects aged 18-64 years, who received 2 doses of placebo at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
  Interventions: Biological: Placebo
- Influenza A (H5N1) >64Y Group (Experimental): Subjects aged > 64 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted vaccine formulations A. B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted
- Placebo >64Y Group (Placebo Comparator): Subjects aged > 64 years, who received 2 doses of placebo at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
  Interventions: Biological: Placebo
- Influenza A (H5N1) Group (Experimental): Pooled group of subjects aged >18 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted vaccine formulations A. B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted
- Placebo Group (Placebo Comparator): Pooled group of subjects aged >18 years, who received 2 doses of placebo at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
  Interventions: Biological: Placebo
- Influenza A (H5N1) 18-60Y Group (Experimental): Subjects aged 18-60 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted vaccine formulations A. B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted
- Placebo 18-60Y Group (Placebo Comparator): Subjects aged 18-60 years, who received 2 doses of placebo at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
  Interventions: Biological: Placebo
- Influenza A (H5N1) >60Y Group (Experimental): Subjects aged >60 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted vaccine formulations A. B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted
- Placebo >60Y Group (Placebo Comparator): Subjects aged > 60 years, who received 2 doses of placebo at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted — Two intramuscular injections at Days 0 and 21.
  Arms: Influenza A (H5N1) 18-60Y Group; Influenza A (H5N1) 18-64Y Group; Influenza A (H5N1) >60Y Group; Influenza A (H5N1) >64Y Group; Influenza A (H5N1) Group
Biological: Placebo — Two intramuscular injections at Days 0 and 21.
  Arms: Placebo 18-60Y Group; Placebo 18-64Y Group; Placebo >60Y Group; Placebo >64Y Group; Placebo Group

SUMMARY:
The purpose of this Phase 3, observer-blind, placebo-controlled, multi-center study is to characterize the immunogenicity & safety of the investigation vaccination regimen of GSK 1557484A vaccine given to adults aged ≥18 years.

ELIGIBILITY:
Inclusion Criteria:

* A male or female 18 years of age or greater at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Among 18 to 49 year old subjects, good general health as established by medical history and clinical examination before entering into the study.
* Among subjects > 49 years of age, stable health status within 1 month prior to enrollment.
* Access to a consistent means of telephone contact.
* Comprehension of the study requirements, ability to comprehend and comply with procedures for collection of short- and long-term safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits.

Exclusion Criteria:

* Evidence of substance abuse or of neurological or psychiatric diagnoses which, even if clinically stable, are deemed by the investigator to render the potential subjectunable/unlikely to provide accurate safety reports.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* An oral temperature ≥37.8º C, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus infection.
* Receipt of systemic glucocorticoids within 1 month of study enrollment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment.
* Any significant disorder of coagulation or treatment with Coumadin derivatives or heparin.
* Administration of any vaccines within 30 days before study enrollment.
* Previous administration of any H5N1 vaccine.
* Use of any investigational or non-registered product or planned participation in another investigational study within 30 days prior to study enrollment, or during the 364 days following the first test article dose. Use of any investigational or non-registered product with immunosuppressive properties is exclusionary at any time during the trial.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrollment or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin test result prior to either vaccination.
* Lactating or nursing.
* Women of child bearing potential who lack a history of reliable contraceptive practices. The provision of this history does NOT replace the requirement to perform, and obtain negative results in pregnancy urine tests prior to treatments.
* Known use of an analgesic or antipyretic medication within 12 hours prior to first treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4561 (Actual)
Dates: Start 2008-01-23; Primary Completion 2008-10-15 (Actual); Study Completion 2009-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (30):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Angelo, Texas
- Canada (10):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Woodstock, Ontario
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint Romuald, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Langley JM, Risi G, Caldwell M, Gilderman L, Berwald B, Fogarty C, Poling T, Riff D, Baron M, Frenette L, Sheldon E, Collins H, Shepard M, Dionne M, Brune D, Ferguson L, Vaughn D, Li P, Fries L. Dose-sparing H5N1 A/Indonesia/05/2005 pre-pandemic influenza vaccine in adults and elderly adults: a phase III, placebo-controlled, randomized study. J Infect Dis. 2011 Jun 15;203(12):1729-38. doi: 10.1093/infdis/jir172. PMID 21606531
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 110464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group
Started | 2304 | 768 | 1118 | 371
Completed | 2242 | 750 | 1101 | 364
Not Completed | 62 | 18 | 17 | 7
Not completed — Adverse Event | 6 | 3 | 2 | 2
Not completed — Other | 51 | 8 | 15 | 5
Not completed — Lost to Follow-up | 5 | 7 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Influenza A (H5N1) 18-64Y Group: Subjects aged 18-64 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, formulations A, B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
- Influenza A (H5N1) >64Y Group: Influenza A (H5N1) >64Y Group Subjects aged > 64 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, formulations A, B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
- Total: Total of all reporting groups
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group | Total
Number analyzed (Participants) | 2304 | 768 | 1118 | 371 | 4561
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (13.64) | 38.7 (13.58) | 71.9 (5.49) | 72.1 (5.41) | 49.5 (19.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1328 | 424 | 621 | 196 | 2569
  Male | 976 | 344 | 497 | 175 | 1992

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects Against A/Indonesia/5/2005 (H5N1)
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination (Day 0) reciprocal HI titer < 1:10 and a post-vaccination (Day 42) reciprocal titer ≥ 1:40, or a pre-vaccination reciprocal HI titer ≥ 1:10 and at least a 4-fold increase in post-vaccination reciprocal titer against A/Indonesia/5/05 virus 21 days after the second dose of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted.
Time Frame: At Day 42 post Dose 1 (Day 42 post Dose 1 = Day 21 post Dose 2)
Population: The analysis was based on the ATP cohort for analysis of immunogenicity, which included all evaluable subjects (meeting all eligibility criteria, complying with the procedures in the protocol, with no elimination criteria during the study) with a complete set of data concerning immunogenicity primary outcome variables available.
Measure: Number; unit: Subjects
Groups:
- Influenza A (H5N1) 18-64Y Group: Subjects aged 18-64 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, formulations A. B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
- Influenza A (H5N1) >64Y Group: Subjects aged > 64 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, formulations A. B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group
Number analyzed (Participants) | 1571 | 76 | 396 | 40
Subjects | 1427 | 1 | 293 | 1

2. Primary Outcome: Number of Seroprotected Subjects Against A/Indonesia/5/2005 (H5N1)
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40.
Time Frame: At Day 0 and Day 42 post Dose 1 (Day 42 post Dose 1 = Day 21 post Dose 2)
Population: as for outcome 1
Measure: Number; unit: Subjects
Groups:
- Influenza A (H5N1) >64Y Group: Subjects aged > 64 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, formulations A, B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group
Number analyzed (Participants) | 1571 | 76 | 396 | 40
Subjects
  Day 0 | 5 | 0 | 9 | 0
  Day 42 | 1467 | 1 | 334 | 1

3. Primary Outcome: Number of Subjects With Any Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During a 7-day follow-up period (i.e., day of vaccination and 6 subsequent days) after each vaccine administration
Population: The analysis was based on the Total Vaccinated cohort, on subjects with symptom sheets completed.
Measure: Number; unit: Subjects
Groups:
- Influenza A (H5N1) Group: Pooled group of subjects aged >18 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, formulations A. B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group | Influenza A (H5N1) Group | Placebo Group
Number analyzed (Participants) | 2267 | 754 | 1109 | 368 | 3376 | 1122
Subjects
  Pain | 2024 | 171 | 784 | 53 | 2808 | 224
  Redness | 181 | 7 | 106 | 1 | 287 | 8
  Swelling | 241 | 7 | 110 | 1 | 351 | 8

4. Primary Outcome: Number of Subjects With Any Solicited General Symptoms.
Description: Assessed solicited general symptoms were fatigue, headache, joint pain at other locations, muscle aches, shivering, sweating and temperature[defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During a 7-day follow-up period (i.e., day of vaccination and 6 subsequent days) after each vaccine administration
Population: The analysis was based on the Total Vaccinated cohort, on subjects with symptom sheets completed.
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group | Influenza A (H5N1) Group | Placebo Group
Number analyzed (Participants) | 2266 | 755 | 1109 | 368 | 3375 | 1123
Subjects
  Fatigue | 890 | 189 | 258 | 64 | 1148 | 253
  Headache | 932 | 249 | 247 | 63 | 1179 | 312
  Joint pain at other location | 645 | 97 | 208 | 39 | 853 | 136
  Muscle aches | 1188 | 175 | 338 | 56 | 1526 | 231
  Shivering | 456 | 87 | 107 | 22 | 563 | 109
  Sweating | 314 | 67 | 48 | 15 | 362 | 109
  Temperature | 121 | 32 | 35 | 6 | 156 | 109

5. Primary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During a 21-day follow-up period for each vaccine administration, as well as overall (Day 0 through Day 84)
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group
Number analyzed (Participants) | 2304 | 768 | 1118 | 371
Subjects
  Unsolicited AEs Days 0-21 | 914 | 289 | 399 | 113
  Unsolicited AEs Days 0-84 | 1017 | 321 | 467 | 130

6. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 through Day 182 and through Day 379.
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group
Number analyzed (Participants) | 2304 | 768 | 1118 | 371
Subjects
  Subjects with SAEs Days 0-182 | 24 | 7 | 43 | 14
  Subjects with SAEs Days 0-379 | 46 | 15 | 65 | 30

7. Primary Outcome: Number of Subjects With Medically Attended Events (MAEs)
Time Frame: From Day 0 through Day 182 and through Day 364.
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group
Number analyzed (Participants) | 2304 | 768 | 1118 | 371
Subjects
  Subjects with MAEs Days 0-182 | 480 | 154 | 298 | 92
  Subjects with MAEs Days 0-379 | 627 | 212 | 400 | 134

8. Secondary Outcome: Number of Subjects With Serum Reciprocal HI Antibodies Against A/Indonesia/5/2005 Equal to or Above (≥) 1:10
Time Frame: At Day 42 post Dose 1 (Day 42 post Dose 1 = Day 21 post Dose 2)
Population: as for outcome 1
Measure: Number; unit: Subjects
Groups:
- Influenza A (H5N1) 18-60Y Group: Subjects aged 18-60 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, formulations A, B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
- Influenza A (H5N1) >60Y Group: Subjects aged >60 years, who received 2 doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, formulations A. B, or C in approximately equal proportions, at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
Arm/Group | Influenza A (H5N1) 18-60Y Group | Placebo 18-60Y Group | Influenza A (H5N1) >60Y Group | Placebo >60Y Group
Number analyzed (Participants) | 1488 | 68 | 479 | 48
Subjects | 1391 | 1 | 410 | 1

9. Secondary Outcome: Number of Subjects With A/Indonesia/5/05 Antibody Titers ≥ 1:10
Time Frame: At Month 6 (Day 182) post Dose 1
Population: The analysis was based on the ATP cohort for analysis of immunogenicity - Month 6, which included all evaluable subjects (meeting all eligibility criteria, complying with the procedures in the protocol, with no elimination criteria during the study) with a complete set of data concerning immunogenicity primary outcome variables available at Month 6
Measure: Number; unit: Subjects
Groups:
- Placebo ˃ 64Y Group: Subjects aged > 64 years, who received 2 doses of placebo at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo ˃ 64Y Group
Number analyzed (Participants) | 366 | 37 | 91 | 19
Subjects | 258 | 2 | 77 | 1

10. Secondary Outcome: Number of Seroconverted Subjects Against A/Indonesia/5/2005 (H5N1)
Description: as for outcome 1
Time Frame: At Month 6 (Day 182) after Dose 1
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group
Number analyzed (Participants) | 366 | 37 | 91 | 19
Subjects | 225 | 1 | 59 | 0

11. Secondary Outcome: Number of Seroprotected Subjects Against A/Indonesia/5/2005 (H5N1)
Time Frame: At Month 6 (Day 182) after Dose 1
Population: as for outcome 9
Measure: Number; unit: Subjects
Groups:
- Placebo >64Y Group: Subjects aged >64 years, who received 2 doses of placebo at Days 0 and 21. The first dose was administered in the deltoid region of the non-dominant arm. The second dose was administered in the deltoid region of the dominant arm.
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group
Number analyzed (Participants) | 366 | 37 | 91 | 19
Subjects | 225 | 1 | 60 | 0

12. Secondary Outcome: Titers for Serum HI Antibodies Against A/Indonesia/5/05 (H5N1)
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was ≥ 1:10.
Time Frame: At Month 6 (Day 182) after Dose 1
Population: The analysis was based on the ATP cohort for analysis of immunogenicity - Month 6, which included all evaluable subjects (meeting all eligibility criteria, complying with the procedures in the protocol, with no elimination criteria during the study) with a complete set of data concerning immunogenicity primary outcome variables at Month 6.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo ˃ 64Y Group
Number analyzed (Participants) | 366 | 37 | 40 | 19
Titers | 36.2 [31.0 to 42.2] | 5.5 [4.8 to 6.5] | 44.8 [33.3 to 60.4] | 5.4 [4.6 to 6.3]

13. Secondary Outcome: Number of Subjects With a Vaccine Response to the Vaccine-homologous Virus and Drift Variant H5N1 Virus, as Assessed by Microneutralization Assays.
Description: Virus antibody response rates were defined as the number of subjects with antibody titers at Day 42 ≥ 4-fold the pre-vaccination antibody titers. The 2 strains assessed were Flu A/Indonesia/5/05 and Flu A/Vietnam/1194/04.
Time Frame: At Day 42 post Dose 1 (Day 42 post Dose 1 = Day 21 post Dose 2)
Population: The analysis was based on the ATP cohort for analysis of immunogenicity, which included all evaluable subjects (meeting all eligibility criteria, complying with the procedures in the protocol, with no elimination criteria during the study) with available data.
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 18-64Y Group | Influenza A (H5N1) >64Y Group
Number analyzed (Participants) | 188 | 46
Subjects
  A/Indonesia/5/05 | 177 | 36
  A/Vietnam/1194/04 | 113 | 12

14. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against A/Vietnam/1194/2004 (H5N1) and A/Indonesia/5/2005 (H5N1) as Assessed by Microneutralization Assays
Description: Titers were expressed as Geometric Mean Titers (GMTs).
Time Frame: At Day 0 and Day 42 post Dose 1 (Day 42 post Dose 1 = Day 21 post Dose 2)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influenza A (H5N1) 18-64Y Group | Influenza A (H5N1) >64Y Group
Number analyzed (Participants) | 188 | 46
Titers
  A/Indonesia/5/05, Day 0 | 22.4 [19.9 to 25.3] | 52.4 [39.2 to 69.8]
  A/Indonesia/5/05, Day 42 | 1450.6 [1266.9 to 1660.9] | 631.1 [444.5 to 896.1]
  A/Vietnam/1194/04, Day 0 | 29.9 [25.7 to 34.9] | 94.4 [68.4 to 130.3]
  A/Vietnam/1194/04, Day 42 | 163.1 [145.6 to 182.8] | 213.4 [165.5 to 275.1]

ADVERSE EVENTS:
Time Frame: SAEs were collected up to Day 182 and up to study end at Day 379. Unsolicited AEs were collected up to Day 20 and up to Day 84. Systematically-assessed symptoms were collected up to Day 6 post vaccination.
Arm/Group | Influenza A (H5N1) 18-64Y Group | Placebo 18-64Y Group | Influenza A (H5N1) >64Y Group | Placebo >64Y Group
Serious Adverse Events (participants affected / at risk) | 24/2304 | 7/768 | 43/1118 | 14/371
Other Adverse Events (participants affected / at risk) | 2087/2304 | 405/768 | 866/1118 | 141/371
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza A (H5N1) 18-64Y Group (N=2304) | Placebo 18-64Y Group (N=768) | Influenza A (H5N1) >64Y Group (N=1118) | Placebo >64Y Group (N=371)
Pneumonia (Infections and infestations) | 1 | 0 | 4 | 2
Myocardial infarction (Cardiac disorders) | 1 | 0 | 3 | 2
Chest pain (General disorders) | 3 | 0 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 3 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 1
Affective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Biopsy liver normal (Surgical and medical procedures) | 0 | 0 | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Caecitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiomegaly (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Carotid artery dissection (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Cholangitis suppurative (Cardiac disorders) | 0 | 0 | 1 | 0
Cholecystitis (Infections and infestations) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis ischaemic (Infections and infestations) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Coronary artery occlusion (Vascular disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enteritis (Infections and infestations) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Gallbladder disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
HIV test positive (Infections and infestations) | 0 | 1 | 0 | 0
Hamartoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hepatitis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Hiatus hernia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hypersensitivity (Psychiatric disorders) | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Vascular disorders) | 1 | 0 | 0 | 0
Left atrial dilatation (Cardiac disorders) | 0 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lymph node cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lymphoma (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0 | 0
Melaena (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Mountain sickness acute (General disorders) | 0 | 0 | 1 | 0
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Nasal septum deviation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pancreatitis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Radiculitis (Nervous system disorders) | 0 | 0 | 1 | 0
Rectal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal tubular acidosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal vessel disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal cord compression (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0
Syncope (General disorders) | 1 | 0 | 0 | 0
Synovial cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tongue carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Toxic nodular goitre (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Transplant rejection (General disorders) | 1 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Urinary retention postoperative (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Influenza A (H5N1) 18-64Y Group (N=2304) | Placebo 18-64Y Group (N=768) | Influenza A (H5N1) >64Y Group (N=1118) | Placebo >64Y Group (N=371)
Pain (General disorders) | 2024/2267 | 171/754 | 784/1109 | 53/368
Redness (General disorders) | 181/2267 | 7/754 | 106/1109 | 1/368
Swelling (General disorders) | 241/2267 | 7/754 | 110/1109 | 1/368
Fatigue (General disorders) | 890/2266 | 189/755 | 258/1109 | 64
Headache (General disorders) | 932/2266 | 249/755 | 247/1109 | 63
Joint pain at other location (General disorders) | 645/2266 | 97/755 | 208/1109 | 39
Muscle aches (General disorders) | 1188/2266 | 175/755 | 338/1109 | 56
Shivering (General disorders) | 456/2266 | 87/755 | 107/1109 | 22
Sweating (General disorders) | 314/2266 | 67/755 | 48/1109 | 15
Temperature (Oral) (General disorders) | 121/2266 | 32/755 | 35/1109 | 6
Nasopharyngitis (Infections and infestations) | 116 | 29 | 40 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 91 | 39 | 34 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.